CLINICAL TRIAL: NCT04754048
Title: A Prospective, Open, Non-comparative, Post-market Clinical Follow-up Investigation to Confirm Safety and Performance of Avance Solo NPWT System in Low to Moderate Exuding Acute (Traumatic Wounds and Flaps and Grafts), as Well as Subacute (e.g., Dehisced Wounds) Wounds
Brief Title: Confirm the Safety and Performance of Avance Solo NPWT System
Acronym: ASOLO-SW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-598655
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Acute Wound; Traumatic Wound; Skin Graft; Skin Flap; Subacute Wound; Dehiscence
Keywords: Negative Pressure Wound Therapy; Post Market Clinical Follow-up

STUDY DESIGN:
Intervention Model Description: Three different patient groups treated with the Avance Solo NPWT System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traumatic wounds (Experimental): Treatment with negative pressure wound therapy.
  Interventions: Device: Avance Solo NPWT System
- Subacute wounds (e.g., dehisced wounds) (Experimental): Treatment with negative pressure wound therapy.
  Interventions: Device: Avance Solo NPWT System
- Flaps and Grafts (Experimental): Treatment with negative pressure wound therapy.
  Interventions: Device: Avance Solo NPWT System

INTERVENTIONS:
Device: Avance Solo NPWT System — Wound treatment with Avance Solo NPWT System for up to 28 days.

SUMMARY:
The primary objective of this post market clinical follow-up (PMCF) investigation is to confirm safety and performance of Avance® Solo NPWT System in low to moderate exuding acute (traumatic wounds and flaps and grafts), as well as subacute (e.g., dehisced wounds) wounds when used in accordance with the Instructions for Use, for up to 28 days.

DETAILED DESCRIPTION:
This investigation is designed as a prospective, open, non-comparative, PMCF investigation to confirm safety and performance of Avance Solo NPWT System in subjects with traumatic wounds (n=34), subacute (e.g., dehisced wounds) wounds (n=34), and flaps and grafts (n=34). This is a multi-center study that will take place in approximately 5 European countries. The eligible subjects will be both in and out patients and all will be treated with Avance Solo NPWT System, for up to 28 days.

Treatment will be stopped if the wound is considered healed, has a high enough percentage of graft take, or enough flap viability by the judgement of the clinicians before the complete treatment time (28 days).

The primary performance endpoint will include assessment of wound progress compared to last visit during a maximum 28 days investigation period. Wound progression is determined by the Investigator and will be assessed at each follow-up visit and measured by three outcomes:

* Deteriorated
* No change
* Improved

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years.
2. Signed written informed consent.
3. Low to moderate exuding acute (traumatic wound, or a flap/graft) or subacute (e.g., dehisced wounds) wounds suitable for single use NPWT according to the investigator´s judgement and Instructions for Use

Exclusion Criteria:

1. Known malignancy in the wound or margins of the wound
2. Untreated and previously confirmed osteomyelitis
3. Non-enteric and unexplored fistulas
4. Necrotic tissue with eschar present
5. Exposed nerves, arteries, veins or organs
6. Exposed anastomotic site
7. Subjects with known allergies/hypersensitivity to product components.
8. Known pregnancy or planning to become pregnant or lactation at the time of study participation.
9. Subjects not suitable for the investigation according to the investigator's judgement and Clinical Investigation Plan and IFU.
10. Participating in other ongoing clinical investigation, or during the past 30 days that may impact the outcome of this investigation based on the judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Change in wound progress | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Wound progress compared to last visit and assessed as:
  * Deteriorated
  * No change
  * Improved

SECONDARY OUTCOMES:
Wound progress | 28 days
  Wound progress compared between baseline and final visit and assessed as:
  * Deteriorated
  * No change
  * Improved
Wound dimension | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Absolute and percentage change in wound area and volume from baseline to all follow-up visits.
Tissue type | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in tissue type (slough, necrotic, granulation or epithelization) from baseline to all follow-up visits.
Exudate | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in exudate amount, nature, and odor using a category scoring system from baseline to all follow-up visits.
  Amount: none, low, moderate, or high
  Nature: serous, fibrinous, serosanguineous, sanguineous, seropurulent, purulent, foul purulent, heamopurulent, or hemorrhagic
  Odor: No odor, slight, moderate, strong, very strong
Peri-wound | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in peri-wound skin condition from baseline to all follow-up visits using the following conditions:
  * Normal
  * Erythematous
  * Oedematous
  * Eczematous
  * Excoriated
  * Macerated
  * Indurated
Pain assessment | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Subject evaluation of pain at Avance Solo dressing removal using Numeric Rating Scale (NRS) at each follow-up visit.
Absorb and transport of exudate | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Clinician evaluation of Avance Solo NPWT System ability to absorb and transport exudate assessed at all follow-up visits
Tissue in-growth | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days) with additional assessments in between when dressing is changed
  Degree of tissue in-growth when Avance Solo foam is utilized at all follow-up visits as well as extra visits.
Trauma | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Proportion of subjects with trauma to the wound site and surrounding skin for Avance Solo Border Dressing and also Avance Solo fixation strips at all follow-up visits
Graft take | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in percentage of graft take and wound epithelization from baseline to all follow-up visits
Flap survival | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in percentage of flap survival from baseline to all follow-up visits
Wear time | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Evaluate Avance Solo NPWT System wear time in days from baseline to all follow-up visits including potential extra visits
Alarms | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Subject evaluation of the Avance Solo NPWT System properties (number of sounding alarms) assessed with a given scale at all follow-up visits
  * 0
  * 1-5
  * 6-10
  * 11-15
  * 16-20
  * More than 20
Product consumption | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Product consumption of the utilized products for the Avance Solo NPWT System, from baseline and final visit using the Avance Solo NPWT System
Quality of life assessment | 28 days
  Subject evaluation of the Avance Solo NPWT system impact of everyday life
Ease of application | Baseline, Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Clinician evaluation of ease of application and removal of the Avance Solo NPWT System using a Numeric Rating Scale (NRS) collected at baseline, and each follow-up visit.
Compliance | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Evaluate the compliance to Avance Solo NPWT System therapy by average number of hours per 24h that the system has not provided treatment since last visit.
Global satisfaction | 28 days
  Evaluate the investigator and subject global satisfaction of the Avance Solo NPWT System in regards to:
  * Very dissatisfied
  * Dissatisfied
  * Neither satisfied or dissatisfied
  * Satisfied
  * Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Beele, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (10):
- Belgium (2):
  - Diensthoofd wondkliniek, UZ Gent, Ghent
  - AZ Delta, Roeselare
- France (2):
  - CHU Montpellier, Montpellier
  - Hôpital Paris St Joseph, Paris
- Germany (2):
  - Franziskus-Krankenhaus Berlin, Berlin
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein Campus Lübeck, Lübeck
- Italy (4):
  - "E. Profili" Civil Hospital, Fabriano
  - Ospedale San Raffaele S.r.l., Milan
  - A.O.U. Citta della Salute e della Scienza di Torino - A.O.U. Molinette San Giovanni Battista, Torino
  - Università dell'Insubria, Varese, Varese

IPD SHARING:
Plan to Share IPD: No